CLINICAL TRIAL: NCT06952361
Title: Evaluation of Alternative Transfusion Triggers in Hemodynamically Stable, Non-Ventilated Cancer Patients: A Prospective Observational Study
Brief Title: Evaluation of Alternative Transfusion Triggers in Hemodynamically Stable, Non-Ventilated Cancer Patients
Status: Completed | Type: Observational
Sponsor: Ardak Arynov (Other)
Responsible Party: Sponsor-Investigator, Ardak Arynov, Head of the Department of Anesthesiology and Intensive Care, Kazakh Institute of Oncology and Radiology, Kazakh Institute of Oncology and Radiology
Organization: Kazakh Institute of Oncology and Radiology (Other)
Other Study IDs: KazIOR-ALTTRANS-2019
Record Dates: First submitted 2025-04-23; First posted 2025-04-30 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-04

CONDITIONS: Anemia; Blood Transfusion; Cancer; Hemoglobin; Alternative Physiological Transfusion Triggers
Keywords: anemia; red blood cell transfusion; physiologic transfusion trigger; alternative transfusion trigger; oxygen extraction ratio; central venous oxygen saturation
MeSH Terms: conditions — Anemia; Neoplasms | interventions — Erythrocyte Transfusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cancer Patients with Anemia Receiving RBC Transfusion: This group includes clinically stable, non-ventilated adult oncology patients with anemia who received red blood cell transfusion at the Kazakh Institute of Oncology and Radiology. All participants were monitored for physiological parameters-including O₂ER, ScvO₂, PvO₂, A-VO₂diff, lactate, and ΔCO₂-before and one hour after transfusion.
  Interventions: Procedure: Red blood cell transfusion

INTERVENTIONS:
Procedure: Red blood cell transfusion — Standard red blood cell transfusion performed as part of routine clinical care. All participants received one or more units of RBCs based on a restrictive hemoglobin threshold. The transfusion protocol was not altered for the purpose of the study.

SUMMARY:
This is a prospective, single-center observational study conducted at the Kazakh Institute of Oncology and Radiology. The study included 107 clinically stable adult patients with cancer who required red blood cell transfusion based on a restrictive hemoglobin threshold. The aim of the study was to evaluate alternative physiological indicators of transfusion need and effectiveness. Measurements included oxygen extraction ratio (O₂ER), central venous oxygen saturation (ScvO₂), partial pressure of oxygen in central venous blood (PvO₂), arterio-venous oxygen difference (A-VO₂diff), lactate, and veno-arterial carbon dioxide difference (ΔCO₂). These parameters were assessed before and one hour after transfusion. For data analysis, patients were stratified into two groups based on their baseline O₂ER (≤35.4% and >35.4%) to evaluate whether higher O₂ER is associated with more pronounced physiological response to transfusion.

ELIGIBILITY:
Inclusion Criteria:

* Adult cancer patients (age 18 years or older)
* Hemodynamically stable
* Not requiring any form of respiratory support
* Presence of a central venous catheter inserted into the superior vena cava

Exclusion Criteria:

* Hemodynamic instability requiring inotropic or vasopressor support
* Active bleeding
* Shock of any etiology
* Patient refusal to participate in the study
* Hematological malignancies
* Age under 18 years
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinically stable, non-ventilated adult oncology patients with anemia who required red blood cell transfusion as part of routine clinical care at the Kazakh Institute of Oncology and Radiology.
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2019-03-08 (Actual); Primary Completion 2021-11-24 (Actual); Study Completion 2021-11-24 (Actual)

PRIMARY OUTCOMES:
Change in Oxygen Extraction Ratio (O₂ER) | Baseline and 1 hour post-transfusion
  Difference in oxygen extraction ratio measured before and one hour after red blood cell transfusion

SECONDARY OUTCOMES:
Change in Partial Pressure of Oxygen in Central Venous Blood (PvO₂) | Baseline and 1 hour post-transfusion
  Difference in PvO₂ measured before and one hour after transfusion
Change in Central Venous Oxygen Saturation (ScvO₂) | Baseline and 1 hour post-transfusion
  Difference in ScvO₂ measured before and one hour after transfusion
Change in Lactate Concentration | Baseline and 1 hour post-transfusion
  Difference in serum lactate measured before and one hour after transfusion
Change in Arterio-Venous Oxygen Difference (A-VO₂diff) | Baseline and 1 hour post-transfusion
  Difference in arteriovenous oxygen difference measured before and one hour after transfusion
Change in Veno-Arterial Carbon Dioxide Difference (ΔCO₂) | Baseline and 1 hour post-transfusion
  Difference in ΔCO₂ measured before and one hour after transfusion

CONTACTS AND LOCATIONS:
Overall Officials: ARDAK A ARYNOV, M.D., Principal Investigator — Department of Anesthesiology and Intensive Care, Kazakh Institute of Oncology and Radiology, Almaty city, Kazakhstan; Evgeni Brotfain, M.D., Professor, Study Chair — Division of Anesthesia and Critical Care, Director of Post Anesthesia Care Unit, Soroka University Medical Center, Ben Gurion University of the Negev, Be'er Sheva, Israel
Locations (1):
- Kazakh Institute of Oncology and Radiology, Almaty, Kazakhstan

IPD SHARING:
Plan to Share IPD: No
The study results will be published in aggregated form only. No individual participant data (IPD) will be shared.

REFERENCES:
- [Derived] Arynov A, Gratz J, Kabon B, Kaidarova D, Satanova A, Brotfain E. Evaluation of alternative transfusion triggers in hemodynamically stable, non-ventilated cancer patients: a prospective observational study. Sci Rep. 2025 Dec 19. doi: 10.1038/s41598-025-32630-6. Online ahead of print. PMID 41419638